CLINICAL TRIAL: NCT06955858
Title: Recombinant Human Thrombopoietin for Autologous Hematopoietic Stem Cell Mobilization in Acute Leukemia: A Single-Arm Prospective Study
Brief Title: Clinical Study of rhTPO in Hematopoietic Stem Cell Mobilization for Autologous Transplantation in Acute Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IIT2025002
Record Dates: First submitted 2025-03-26; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic Stem Cell Mobilization
Keywords: Recombinant Human Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The group of rhTPO (Experimental)
  Interventions: Drug: Recombinant Human Thrombopoietin（rhTPO）

INTERVENTIONS:
Drug: Recombinant Human Thrombopoietin（rhTPO） — G-CSF will be administered at a dose of 10 μg/kg/day subcutaneously for 7-10 days post-chemotherapy.
  rhTPO is started on the same day as G-CSF at 300 U/kg/d and injected subcutaneously until the stem cell collection was completed.

SUMMARY:
Evaluation of the efficacy and safety of recombinant human thrombopoietin (rhTPO) at 300 U/kg/day for hematopoietic stem cell mobilization in autologous transplantation among acute leukemia patients

ELIGIBILITY:
Inclusion Criteria:

1. Age 18～65 years, regardless of gender.
2. Histopathologically confirmed acute leukemia with immunohistochemical validation
3. Sustained complete hematologic remission with documented minimal residual disease (MRD) negativity.
4. Eastern Cooperative Oncology Group (ECOG) performance status smaller than 2 and a life expectancy of more than 6 months
5. No active infectious disease; no severe organ failure.
6. Willingness to participate with written informed consent for study enrollment.

Exclusion Criteria:

1. Liver dysfunction (alanine aminotransferase or bilirubin greater than two times the normal upper limit).
2. Renal dysfunction (creatinine or urea higher than 1.5 times the normal upper limit).
3. Any disease that could put patients at high risk, including but not limited to unstable cardiac disease, uncontrolled atrial fibrillation or hypertension, severe diabetic retinopathy
4. rhTPO aller- gies.
5. Severe prior thrombosis-event.
6. History of other malignancy, unless cured for more than 3 years
7. Pregnant or lactating women
8. Severe infectious disease (uncured tuberculosis, pulmonary aspergillosis)
9. Epilepsia, dementia or any mental disease requiring treatment.
10. Other conditions deemed inappropriate for study participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
total CD34+ cell count | two weeks
  Median total number of CD34+ cells collected

SECONDARY OUTCOMES:
the proportion of patients collecting more than or equal to 2*10^6 CD34+ cells/kg | two weeks
the proportion of patients collecting more than or equal to 5*10^6 CD34+ cells/kg | two weeks
total mononuclear cell count | two weeks
  Median total number of mononuclear cells collected
time of platelet engraftment | eight weeks
  defined as platelet count >20×109 platelets/L for seven consecutive days without platelet transfusion
time of neutrophil engraftment | four weeks
  defined as the absolute value of neutrophils >0.5×109 cells/L for three consecutive days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China